CLINICAL TRIAL: NCT06723561
Title: Low Dose Naltrexone in the Treatment of Central Neuropathic Pain After Traumatic Spinal Cord Injury: A Pilot Study
Brief Title: Treating Central Neuropathic Pain With Low Dose Naltrexone for People With Spinal Cord Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Chen Cui, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 51429
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Central Neuropathic Pain; Spinal Cord Injury
Keywords: Central Neuropathic Pain; CNP; Spinal Cord Injury; SCI; Naltrexone; Low Dose Naltrexone; LDN
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low Dose Naltrexone (Experimental): Daily dose of 4.5mg of naltrexone
  Interventions: Drug: 4.5mg daily dose of naltrexone

INTERVENTIONS:
Drug: 4.5mg daily dose of naltrexone — Study subjects will take a daily 4.5mg dose of naltrexone.

SUMMARY:
The goal of this pilot clinical trial is to find out how well low dose naltrexone works for people with pain due to spinal cord injury. The main questions it aims to answer are: will low dose naltrexone reduce pain, and increase the quality of life for people with central neuropathic pain due to spinal cord injury.

Hypothesis 1: LDN will decrease the severity of CNP in adult patients with SCI as measured by the Neuropathic Pain Scale (NPS) Hypothesis 2: LDN will improve quality of life of patients with SCI as measured by various validated clinical tools

There is no comparison group. This study is being completed to give investigators more information for how to best run a larger clinical trial.

Participants will be asked to take an oral dose of 4.5mg of naltrexone, daily, for 12 weeks.

DETAILED DESCRIPTION:
This study is being completed to provide the first evidence that low dose naltrexone may be able to lower pain and improve quality of life for people with pain due to spinal cord injury. Data from this study will be used to plan a larger, randomized control trial. If eligible, participants will take a daily low dose naltrexone pill (4.5mg) by mouth for 12 weeks. Study participants will keep a daily medicine log and a daily sleep log. The study team will check in regularly (virtual visits) with the participants and give questionnaires verbally.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a traumatic cervical or thoracic spinal cord injury
2. Age ≥18
3. >6 months from time of injury
4. Central neuropathic pain related to SCI, based on evaluation of a Physical Medicine & Rehabilitation Physician
5. DN4 questionnaire ≥ 4
6. English speaking

Exclusion Criteria:

1. Adjustment in pain medications within the previous month
2. Chronic opioid treatment
3. Current treatment with naltrexone or other opioid antagonist
4. Allergy to naltrexone
5. Central neuropathic pain attributed to other etiology
6. Neuropathic pain attributed to the peripheral nervous system
7. PHQ9 ≥15 indicating moderately severe or severe depressive symptoms
8. Documented traumatic brain injury that would affect study participation, in the opinion of the investigator
9. Scheduled elective surgery during the duration of the study
10. Pregnant or breastfeeding
11. Illicit substance use per Wisconsin law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate LDN in the treatment of CNP after SCI | From enrollment to the end of treatment at 12 weeks
  Generate initial data to calculate an effect size of LDN in the treatment of CNP in SCI. This will be utilized to plan a randomized control trial and submit for extramural funding.

SECONDARY OUTCOMES:
Evaluate improvement in quality of life using the Average Daily Pain Score (ADPS). | From enrollment to the end of treatment at 12 weeks
  Evaluate improvement in quality of life using the Average Daily Pain Score (ADPS). Participants report a pain score from 0 - no pain, to 10 - the worst pain possible. A lower score is a better outcome.
Evaluate improvement in quality of life using Daily Sleep Interference Scale (DSIS) | From enrollment to the end of treatment at 12 weeks
  Evaluate improvement in quality of life using Daily Sleep Interference Scale (DSIS). Participants report a score between 0 - Pain did not interfere with sleep to 10 - Pain completely interfered with sleep, or was unable to sleep due to pain. A lower score is a better outcome.
Evaluate improvement in quality of life using the Patient Global Impression of Change (PGIC) | From enrollment to the end of treatment at 12 weeks
  Evaluate improvement in quality of life using the Patient Global Impression of Change (PGIC) . Participants report a pain score of overall change in status from 1 - Very much improved to 7 - Very much worse. A lower score is a better outcome.
Evaluate improvement in quality of life using the Neuropathic Pain Scale (NPS). | From enrollment to the end of treatment at 12 weeks
  Evaluate improvement in quality of life using the Neuropathic Pain Scale (NPS). Participants report a pain score from 0 - no pain, to 10 - the worst pain possible. A lower score is a better outcome.
Evaluate improvement in quality of life using the Spinal Cord Injury Quality of Life Pain Interference Scale (SCI-QOL). | From enrollment to the end of treatment at 12 weeks
  Evaluate improvement in quality of life using the Spinal Cord Injury Quality of Life Pain Interference Scale (SCI-QOL). Participants respond to a series of questions about how much pain due to spinal cord injury affects quality of life answering from 1 - Not at all, to 7 - Very much. A lower score is a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study. Data will be used to plan a larger randomized control trial.